CLINICAL TRIAL: NCT04131725
Title: Cardiac Function Monitoring System Evaluation
Brief Title: Cardiac Function Non-Invasive Monitoring System Evaluation Trial
Status: Completed | Type: Observational
Sponsor: Sensydia Corporation (Industry)
Collaborators: University of Pittsburgh Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: CPS_002_2019
Record Dates: First submitted 2019-10-14; First posted 2019-10-18 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cardiac Function Monitoring: Subjects will wear Cardiac Performance System (CPS) non-invasive device for brief periods during procedures including assessment by Pulmonary Artery Catheter (PAC) methods.
  Interventions: Device: Cardiac Performance System (NSR)

INTERVENTIONS:
Device: Cardiac Performance System (NSR) — Device: Cardiac Performance System Participants will be asked to wear the Cardiac Performance System, a non-invasive sensor device on their upper abdomen. The Cardiac Performance System monitoring device will continuously monitor cardiac function. The device will be worn at the time when Pulmonary Artery Catheter procedures are conducted.

SUMMARY:
Non-significant risk device study to conduct evaluation of the performance of new device for monitoring of cardiac function (based on previous iterations 510(k) 173156)

DETAILED DESCRIPTION:
Non-significant risk device study to conduct evaluation of the performance of new device for monitoring of cardiac function (based on previous iterations 510(k) 173156)

ELIGIBILITY:
Inclusion Criteria:

* Adults of age 18 or older

Exclusion Criteria:

* Subjects with wounds or surgical incisions at the site of sensor placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for Pulmonary Artery Catheter procedure
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Cardiac Performance System electronic data for Cardiac Output | 60 minutes during Pulmonary Artery Catheter procedure
  Cardiac function metric measurement including Cardiac Output to report in L/m.
Cardiac Performance System electronic data for Pulmonary Artery Pressure | 60 minutes during Pulmonary Artery Catheter procedure
  Cardiac function metric measurement including Pulmonary Artery Pressure to report in mmHg.
Cardiac Performance System electronic data for Pulmonary Artery Wedge Pressure | 60 minutes during Pulmonary Artery Catheter procedure
  Cardiac function metric measurement including Pulmonary Artery Wedge Pressure to report in mmHg.
Pulmonary Artery Catheter electronic data for Cardiac Output | 60 minutes during Pulmonary Artery Catheter procedure
  Cardiac function metric measurement including Cardiac Output to report in L/m.
Pulmonary Artery Catheter electronic data for Pulmonary Artery Pressure | 60 minutes during Pulmonary Artery Catheter procedure
  Cardiac function metric measurement including Pulmonary Artery Pressure to report in mmHg.
Pulmonary Artery Catheter electronic data for Pulmonary Artery Wedge Pressure | 60 minutes during Pulmonary Artery Catheter procedure
  Cardiac function metric measurement including Pulmonary Artery Wedge Pressure to report in mmHg.
Echocardiography electronic data for Ejection Fraction | 15 minutes at a time prior to or after Pulmonary Artery Catheter procedure
  Cardiac function measurement including left ventricle ejection fraction to report in percentage.

CONTACTS AND LOCATIONS:
Overall Officials: William Kaiser, PhD, Principal Investigator — Sensydia Corporation
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No